CLINICAL TRIAL: NCT05686356
Title: A Novel 4-month Pan-TB Regimen Targeting Both Host and Microbe (panTB-HM)
Brief Title: A Pan-TB Regimen Targeting Host and Microbe
Acronym: panTB-HM
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The Aurum Institute NPC (Other)
Collaborators: Ludwig-Maximilians - University of Munich (Other); Stichting Katholieke Universiteit (Other); Wits Health Consortium (Pty) Ltd (Other); Instituto Nacional de Saúde, Mozambique (Other Government); National Institute for Medical Research, Tanzania (Other Government); University of Stellenbosch (Other); Sequella, Inc. (Industry); Global Alliance for TB Drug Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AUR1-1-312; 24206 (Registry Identifier: Pan African Clinical Trials Registry (PACTR)); 6986 (Registry Identifier: South African Clinical Trials Registry (SANCTR)); RIA2019AMR-2647 (Other Grant/Funding Number: EDCTP)
Record Dates: First submitted 2022-12-18; First posted 2023-01-17 (Actual); Last update posted 2025-05-28 (Actual); Status verified 2025-05

CONDITIONS: Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — PNU-100480; Acetylcysteine; pretomanid; bedaquiline

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Arm 1 (S1200BP) (Experimental): Sutezolid 1200mg QD plus bedaquiline and pretomanid for 4 months
  Interventions: Drug: Sutezolid; Drug: Pretomanid; Drug: Bedaquiline
- Arm 2 (S1600BP) (Experimental): Sutezolid 1600mg QD plus bedaquiline and pretomanid for 4 months
  Interventions: Drug: Sutezolid; Drug: Pretomanid; Drug: Bedaquiline
- Arm 3 (S1600BPN) (Experimental): Sutezolid 1600mg QD plus bedaquiline pretomanid and N-acetyl cysteine for 4 months
  Interventions: Drug: Sutezolid; Drug: N-acetyl cysteine; Drug: Pretomanid; Drug: Bedaquiline
- Arm 4 (HRZE) (Active Comparator): Rifafour (2HRZE/4HR)
  Interventions: Combination Product: Rifafour

INTERVENTIONS:
Drug: Sutezolid — Sutezolid will be given at a dose of 1200mg QD in arm 1 and at a dose of 1600mg QD in arms 2 and 3.
  Arms: Arm 1 (S1200BP); Arm 2 (S1600BP); Arm 3 (S1600BPN)
Drug: N-acetyl cysteine — NAC will be given at a dose of 1800 mg BID in arm 3
  Other Names: NAC
  Arms: Arm 3 (S1600BPN)
Drug: Pretomanid — Pretomanid will be given at its approved dose
  Arms: Arm 1 (S1200BP); Arm 2 (S1600BP); Arm 3 (S1600BPN)
Drug: Bedaquiline — Bedaquiline will be given at its approved dose
  Arms: Arm 1 (S1200BP); Arm 2 (S1600BP); Arm 3 (S1600BPN)
Combination Product: Rifafour — Fixed dose combination tablets for TB treatment will be given at approved doses
  Arms: Arm 4 (HRZE)

SUMMARY:
This project will develop the first regimen meeting WHO criteria for a pan-TB indication, ie, not requiring knowledge of RIF susceptibility. The regimen will test sutezolid at 2 dose levels, with the approved anti-TB drugs bedaquiline and pretomanid, in a phase 2c trial. It will also test whether the addition of N-acetylcysteine (NAC), a re-purposed host-directed WHO essential medicine, can protect the lung and liver against oxidative damage, preserve lung function, and accelerate the eradication of MTB infection by replenishing glutathione (GSH).

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 to 65 years
2. Willing and able to provide signed written consent prior to undertaking any trial-related procedures, or, in the case of illiteracy, witnessed oral consent
3. Body weight (in light clothing without shoes) between 30 and 90 kg.
4. Radiographic evidence of pulmonary tuberculosis
5. Positive Xpert TB/RIF (original or Ultra) for MTB
6. RIF susceptibility diagnosed by Xpert TB/RIF, with subsequent culture confirmation
7. If sexually active, willing to use an effective contraceptive method for the duration of tuberculosis treatment
8. HIV-1 seronegative, or if HIV-1 seropositive, CD4 T cell count ≥100/µl and either receiving ART or willing to start ART during study participation
9. SARS-CoV-2 PCR or antigen test negative, or if positive, either fully vaccinated against Covid-19 or with D-dimer <0.8 ug/ml
10. Willing to adhere to a diet excluding tyramine-rich foods (certain mold-ripened cheeses and cured meats), and to avoid eating grapefruits and pomelos

Exclusion Criteria:

1. Any condition for which participation in the trial, as judged by the investigator, could compromise the well-being of the subject or prevent, limit or confound protocol specified assessments
2. Current or imminent (within 24 hr) treatment for malaria.
3. Pregnant or nursing
4. Is critically ill, and in the judgment of the investigator has a diagnosis likely to result in death during the trial or the follow-up period.
5. TB meningitis or spondylitis, or other forms of severe tuberculosis with high risk of a poor outcome as judged by the investigator.
6. History of allergy or hypersensitivity to any of the trial therapies or related substances.
7. Having participated in other clinical trials with investigational agents within 8 weeks prior to trial start or currently enrolled in an investigational trial.
8. Prior TB treatment in the preceding 6 months
9. Angina pectoris requiring treatment with nitroglycerin or other nitrates
10. Cardiac arrhythmia requiring medication, or any clinically significant ECG abnormality, in the opinion of the investigator
11. History of unstable Diabetes Mellitus requiring hospitalization for hyper- or hypo-glycaemia within the past year prior to start of screening.
12. Use of systemic corticosteroids within the past 28 days.
13. Patients requiring treatment with medications not compatible with rifampin, such as HIV-1 protease inhibitors
14. Patients requiring treatment with antidepressants, including MAO inhibitors and SSRIs.
15. Subjects with any of the following abnormal laboratory values:

    1. HBsAg positive
    2. creatinine >2 mg/dL
    3. hemoglobin <8 g/dL
    4. platelets <100x109 cells/L
    5. serum potassium <3.5 mM/L
    6. alanine aminotransferase (ALT) ≥2.0 x ULN
    7. alkaline phosphatase (AP) >5.0 x ULN
    8. total bilirubin >1.5 mg/dL
    9. random blood glucose >200 mg/dL

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Estimated)
Dates: Start 2023-07-28 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients achieving durable (non-relapsing) cure | Assessed after 1 year of post-treatment follow-up

SECONDARY OUTCOMES:
The proportion of subjects with TE ALT increases, graded according to severity | From day 1 through 4 weeks post end-of-treatment
The proportion of subjects with TE increases in transaminases and bilirubin meeting Hy's criteria for serious liver injury | From day 1 through 4 weeks post end-of-treatment
The proportion of subjects with TE AEs, according to seriousness | From day 1 through 4 weeks post end-of-treatment
The number of TE AEs per treatment arm, according to seriousness | From day 1 through 4 weeks post end-of-treatment
The proportion of subjects requiring temporary or permanent treatment discontinuation due to safety or tolerability concerns | From day 1 through 4 weeks post end-of-treatment
FEV1 and FVC at 1, 2, 6, and 18 months after initiation of treatment | 1, 2, 6, and 18 months after initiation of treatment
FEV1 and FVC slope during 6 and 18 months after initiation of treatment | 6 and 18 months after initiation of treatment
FEV1/FVC ratio at 1, 2, 6, and 18 months after initiation of treatment | 1, 2, 6, and 18 months after initiation of treatment
The proportion of subjects with sputum cultures showing growth of MTB at 1, 2, 3, and 4 months after initiation of treatment | 1, 2, 3, and 4 months after initiation of treatment
The hazard ratio for stable culture conversion through the 4th month of treatment | through the 4th month of treatment
The proportion of subjects with treatment failure | More than 1 specimen showing growth of MTB during the final 6 weeks of treatment
The proportion of subjects with relapse | At week 72 for the control arm and at week 64 for the experimental arms

OTHER OUTCOMES:
The proportion of subjects with non-TB cardiac or pulmonary AEs during the 18 months after TB diagnosis, according to seriousness. | During the 18 months after TB diagnosis
The plasma concentration (AUC) of sutezolid and its main metabolite | Month 1
The plasma concentration (Cmax and Cmin) of sutezolid and its main metabolite | Month 1
The plasma concentration (T>MIC) of sutezolid and its main metabolite | Month 1

CONTACTS AND LOCATIONS:
Overall Officials: Professor Robert Wallis, MD, Principal Investigator — The Aurum Institute NPC
Locations (8):
- Instituto Nacional de Saúde, Maputo, Mozambique
- South Africa (6):
  - Clinical HIV Research Unit, Durban, Durban
  - Clinical HIV Research Unit, Johannesburg, Gauteng
  - The Aurum Institute: Tembisa Clinical Research Centre, Tembisa, Gauteng
  - The Aurum Institute, Gavin J Churchyard Legacy Centre (Klerksdorp Clinical Research Centre), Klerksdorp, Klerksdorp
  - The Aurum Institute, Rustenburg Clinical Research Centre, Rustenburg, North West Provice
  - TASK Eden, George, Western Cape
- NIMR-Mbeya Medical Research Centre, Mbeya, Tanzania

IPD SHARING:
Plan to Share IPD: Yes